CLINICAL TRIAL: NCT05937230
Title: Long-Term Performance of Drug-coated Balloons and Drug-eluting Stents in Diabetic Patients: a Real-world, Prospective Study
Brief Title: Drug-coated Balloons and Drug-eluting Stents in Diabetic Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Ling Tao, MD, PhD, Professor in Cardiology, Director of the department of Cardiology, Xijing Hospital
Other Study IDs: CAGE-FREE DM registry
Record Dates: First submitted 2023-06-29; First posted 2023-07-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Coronary Heart Disease; Angioplasty, Balloon
Keywords: Drug-eluting stents; Drug-coated balloons; Diabetic; De-novo; In-stent stenosis; All-comers
MeSH Terms: conditions — Coronary Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Drug-coated balloon: Paclitaxel coated balloon
  Interventions: Device: Drug-coated balloon
- Drug-eluting stent: Second-generation eluting stents
  Interventions: Device: Drug-eluting stents

INTERVENTIONS:
Device: Drug-coated balloon — Paclitaxel is a pharmacologically active substance for anti-neointima.
  Groups: Drug-coated balloon
Device: Drug-eluting stents — Drug-eluting stent is composed of a metal stent, primer, and drug coating.
  Groups: Drug-eluting stent

SUMMARY:
Drug-eluting stents (DES) have long been recommended as the default device for patients undergoing percutaneous coronary intervention (PCI). Drug-Coated Balloon (DCB) angioplasty is similar to plain old balloon angioplasty procedurally, but there is an anti-proliferative medication paclitaxel-coated on the balloon.

DCB angioplasty has the following advantages compared to DES implantation: Firstly, the drug in DCB is uniformly distributed and released, whereas the drug release of DES via the stent platform is uneven -85% of the vascular wall is not covered by the stent strut. Secondly, there is no alloy in the vessel after DCB angioplasty, while the coronary stent platform and polymer might cause temporal or persistent inflammatory response leading to intimal hyperplasia. Finally, there is no metal cage restraining vessel motion after DCB, and the physiological function of coronary arteries would be maintained.

Currently, DCB constitutes an important treatment option in ISR, which is endorsed by the 2018 European Society of Cardiology Guidelines on myocardial revascularization. In addition, some interventional cardiologist has also applied DCB in de novo lesions in their clinical practice.

Diabetes is associated with worse outcomes after coronary revascularization and has been identified as an independent predictor of adverse events in patients with cardiovascular disease. Although some small sample size RCTs and observational studies have suggested that the clinical prognosis of DCB is non-inferior to the drug-eluting stent (DES), there is still a lack of evidence comparing the DCB versus DES for de novo or ISR coronary lesions in diabetic patients. The current study aims to compare the long-term efficacy of DCB to DES in de novo or ISR coronary lesions in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diabetes mellitus
2. Received PCI by a drug-coated balloons only strategy or drug-eluting stents only strategy

Exclusion Criteria:

1. Under the age of 18
2. Unable to give informed consent
3. Currently participating in another trial or participants unable to comply to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All diabetic patients who received PCI with one or more drug-coated balloons only or drug-eluting stents only to treat ISR or de novo lesions
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Device-oriented Composite Endpoint (DoCE) | 24 months
  DoCE is a composite clinical endpoint of Cardiac cause death, Target vessel myocardial infarction (TV-MI), and clinically indicated target lesion revascularization (CI-TLR).

OTHER OUTCOMES:
POCE | 1 month, and 1, 2, 3, 5, 7, 10 years
  POCE is a composite clinical endpoint of all-cause death, any stroke, non-fatal myocardial infarction (MI), any revascularization
All-cause death | 1 month, and 1, 2, 3, 5, 7, 10 years
  Rates of individual components of PoCE
Non-fatal myocardial infarction (MI) | 1 month, and 1, 2, 3, 5, 7, 10 years
  Rates of individual components of PoCE
Any stroke | 1 month, and 1, 2, 3, 5, 7, 10 years
  Rates of individual components of PoCE
Any revascularization | 1 month, and 1, 2, 3, 5, 7, 10 years
  Rates of individual components of PoCE
Device-oriented Composite Endpoint (DoCE) | 1 month, and 1, 2, 3, 5, 7, 10 years
  Rates of the DoCE beside the time point of primary endpoint
Cardiac cause death | 1 month, and 1, 2, 3, 5, 7, 10 years
  Rates of individual components of the DoCE
Target vessel myocardial infarction (TV-MI) | 1 month, and 1, 2, 3, 5, 7, 10 years
  Rates of individual components of the DoCE
Clinically indicated target lesion revascularization (CI-TLR) | 1 month, and 1, 2, 3, 5, 7, 10 years
  Rates of individual components of the DoCE
Target vessel failure (TVF) | 1 month, and 1, 2, 3, 5, 7, 10 years
  Target vessel failure, defined as cardiovascular death, TV MI and clinically-indicated target vessel revascularisation

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, MD, Ph.D., Study Chair — Xijing Hospital; Chao Gao, MD, Ph.D., Study Chair — Xijing Hospital
Locations (1):
- Ling Tao, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No